CLINICAL TRIAL: NCT01217749
Title: An Open-label, Phase 1b/2, Safety and Efficacy Study of the Bruton's Tyrosine Kinase (Btk) Inhibitor, PCI-32765, and Ofatumumab in Subjects With Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma and Prolymphocytic Leukemia
Brief Title: Efficacy and Safety Study of PCI-32765 Combine With Ofatumumab in CLL
Acronym: PCYC-1109-CA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1109-CA; PCI-32765 (Other: Pharmacyclics)
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Results first posted 2015-04-16 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-05

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Prolymphocyctic Leukemia; Richter's Transformation
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): In Group 1, PCI-32765 420 mg PO was administered daily for 1 cycle (28 days) before the start of ofatumumab IV dosing
  Interventions: Drug: PCI-32765; Drug: ofatumumab
- Group 2 (Experimental): In Group 2, PCI-32765 420 mg PO daily was initiated concomitantly with ofatumumab IV (PCI-32765 initiated on Day 2 of Cycle 1)
  Interventions: Drug: PCI-32765; Drug: ofatumumab
- Group 3 (Experimental): In Group 3, two cycles of ofatumumab IV were administered prior to the start of PCI-32765 420 mg PO daily
  Interventions: Drug: PCI-32765; Drug: ofatumumab

INTERVENTIONS:
Drug: PCI-32765 — 420 mg PO daily
  Other Names: ibrutinib
Drug: ofatumumab — per package insert as an IV infusion
  Other Names: Arzerra

SUMMARY:
The purpose of this study is to determine the efficacy and safety of a fixed-dose, daily regimen of orally administered PCI-32765 combined with ofatumumab in subjects with relapsed/refractory CLL/SLL and related diseases

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histologically confirmed chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL), prolymphocytic leukemia (PLL), or Richter's transformation arising out of CLL/SLL as defined by WHO classification of hematopoietic neoplasms and satisfying ≥ 1 of the following conditions:

   * Progressive splenomegaly and/or lymphadenopathy identified by physical examination or radiographic studies
   * Anemia (<11 g/dL) or thrombocytopenia (<100,000/μL) due to bone marrow involvement
   * Presence of unintentional weight loss > 10% over the preceding 6 months
   * NCI CTCAE Grade 2 or 3 fatigue
   * Fevers > 100.5 degree or night sweats for > 2 weeks without evidence of infection
   * Progressive lymphocytosis with an increase of > 50% over a 2 month period or an anticipated doubling time of < 6 months
   * Need for cytoreduction prior to stem cell transplant
2. Subjects must have failed ≥ 2 prior therapies for CLL including a nucleoside analog or ≥ 2 prior therapies not including nucleoside analog if there is a contraindication to such therapy
3. 10% expression of CD20 on CLL/SLL cells
4. ECOG performance status ≤ 2
5. Life expectancy ≥ 12 weeks
6. Subjects must have organ and marrow function as defined below:

   * Absolute neutrophil count (ANC) ≥ 1000/µL in the absence of bone marrow involvement
   * Platelets ≥ 30,000/μL in the absence of bone marrow involvement
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal unless due to Gilbert's disease
   * AST (SGOT) ≤ 2.5 x institutional upper limit of normal unless due to infiltration of the liver
   * Creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 50 mL/min
7. No history of prior exposure to ofatumumab
8. Age ≥ 18 years
9. Body weight ≥ 40 kg

Exclusion Criteria:

1. A life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of PCI-32765 PO, or put the study outcomes at undue risk
2. Significant cardiovascular disease
3. Any condition which could interfere with the absorption or metabolism of PCI-32765 including unable to swallow capsules, malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction
4. Known history of Human Immunodeficiency Virus (HIV) or active infection with Hepatitis C Virus (HCV) or Hepatitis B Virus (HBV) or any uncontrolled active systemic infection
5. Any anticancer immunotherapy, chemotherapy, radiotherapy, or experimental therapy within 4 weeks before first dose of study drug. Corticosteroids for disease-related symptoms are allowed provided 1 week washout occurs
6. Active central nervous system (CNS) involvement by lymphoma
7. Major surgery within 4 weeks before first dose of study drug
8. Lactating or pregnant
9. Known moderate to severe chronic obstructive pulmonary disease (COPD)
10. History of prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for at least 2 years or which will not limit survival to < 2 years
11. History of Grade ≥ 2 toxicity continuing from prior anticancer therapy including radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2010-12; Primary Completion 2013-06 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Jaglowski, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Derived] Fraietta JA, Beckwith KA, Patel PR, Ruella M, Zheng Z, Barrett DM, Lacey SF, Melenhorst JJ, McGettigan SE, Cook DR, Zhang C, Xu J, Do P, Hulitt J, Kudchodkar SB, Cogdill AP, Gill S, Porter DL, Woyach JA, Long M, Johnson AJ, Maddocks K, Muthusamy N, Levine BL, June CH, Byrd JC, Maus MV. Ibrutinib enhances chimeric antigen receptor T-cell engraftment and efficacy in leukemia. Blood. 2016 Mar 3;127(9):1117-27. doi: 10.1182/blood-2015-11-679134. Epub 2016 Jan 26. PMID 26813675
- [Derived] Maddocks KJ, Ruppert AS, Lozanski G, Heerema NA, Zhao W, Abruzzo L, Lozanski A, Davis M, Gordon A, Smith LL, Mantel R, Jones JA, Flynn JM, Jaglowski SM, Andritsos LA, Awan F, Blum KA, Grever MR, Johnson AJ, Byrd JC, Woyach JA. Etiology of Ibrutinib Therapy Discontinuation and Outcomes in Patients With Chronic Lymphocytic Leukemia. JAMA Oncol. 2015 Apr;1(1):80-7. doi: 10.1001/jamaoncol.2014.218. PMID 26182309
- [Derived] Jaglowski SM, Jones JA, Nagar V, Flynn JM, Andritsos LA, Maddocks KJ, Woyach JA, Blum KA, Grever MR, Smucker K, Ruppert AS, Heerema NA, Lozanski G, Stefanos M, Munneke B, West JS, Neuenburg JK, James DF, Hall N, Johnson AJ, Byrd JC. Safety and activity of BTK inhibitor ibrutinib combined with ofatumumab in chronic lymphocytic leukemia: a phase 1b/2 study. Blood. 2015 Aug 13;126(7):842-50. doi: 10.1182/blood-2014-12-617522. Epub 2015 Jun 26. PMID 26116658
- [Derived] Dubovsky JA, Beckwith KA, Natarajan G, Woyach JA, Jaglowski S, Zhong Y, Hessler JD, Liu TM, Chang BY, Larkin KM, Stefanovski MR, Chappell DL, Frissora FW, Smith LL, Smucker KA, Flynn JM, Jones JA, Andritsos LA, Maddocks K, Lehman AM, Furman R, Sharman J, Mishra A, Caligiuri MA, Satoskar AR, Buggy JJ, Muthusamy N, Johnson AJ, Byrd JC. Ibrutinib is an irreversible molecular inhibitor of ITK driving a Th1-selective pressure in T lymphocytes. Blood. 2013 Oct 10;122(15):2539-49. doi: 10.1182/blood-2013-06-507947. Epub 2013 Jul 25. PMID 23886836
- See also: www.pharmacyclics.com — http://Pharmacyclics.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3
Started | 27 | 20 | 24
Completed | 24 | 17 | 22
Not Completed | 3 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 27 | 20 | 24 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 15 | 40
  >=65 years | 14 | 8 | 9 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 7 | 22
  Male | 19 | 13 | 17 | 49
Region of Enrollment [Number; unit: participants]
  United States | 27 | 20 | 24 | 71

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Response
Description: The primary endpoint for the study was overall response rate (ORR), defined as the proportion of participants who achieved a best overall response of complete response (CR), CR with incomplete blood count recovery (Cri), or partial response (PR), according to the guidelines from the International Workshop on Chronic Lymphocytic Leukemia (IWCLL1) published in 2008 for CLL participants and International Working Group for non-Hodgkin's lymphoma (IWG NHL) 2007 criteria for SLL participants, with the modification that treatment-related lymphocytosis will not be considered progressive disease, as evaluated by the investigators. Assessment of disease is based on radiological exams, physical exam, hematological evaluations and, when appropriate, bone marrow results.
Time Frame: The median follow-up time on study for all treated participants is 12.5 (range 0.5-19.6) months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Group 1: In Group 1, PCI-32765 420 mg PO administered daily for 1 cycle (28 days) before the start of ofatumumab IV dosing
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 27 | 20 | 24
percentage of participants | 92.6 [75.7 to 99.1] | 80.0 [56.3 to 94.3] | 70.8 [48.9 to 87.4]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: Number of participants who had experienced at least one treatment emergent AE
Time Frame: From first dose of study treatment to within 30 days of last dose or until study closure
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 27 | 20 | 24
participants | 27 | 20 | 24

3. Secondary Outcome: Progression Free Survival (PFS) at 12 Months
Description: Progressive disease for CLL (Hallek) is characterized by ≥1 of the following:
  * Appearance of any new lesion, eg lymph nodes (> 1.5 cm), de novo hepatomegaly or splenomegaly, or other organ infiltrates
  * Increase of ≥50%
    * in longest diameter of any previous site
    * in hepatomegaly or splenomegaly
    * in blood lymphocytes with ≥5x109/L B cells with enlarging lymph node, liver, or spleen
  Progressive disease for B cell lymphoma (Cheson) is characterized by any new lesion or increase by ≥ 50% of previously involved sites from nadir:
  * Appearance of a new lesion(s) >1.5 cm in any axis, ≥ 50% increase in the SPD of >1 node, or ≥50% increase in longest diameter of a previously identified node >1 cm in short axis
  * Lesions PET+ if FDG-avid lymphoma or PET+ before therapy
  * 50% increase from nadir in the SPD of any liver or spleen lesions
  * New or recurrent BM involvement
  * Increase of ≥50% in blood lymphocytes with ≥5x109/L B cells within enlarging lymph node, liver, or spleen
Time Frame: From first dose of study treatment until disease progression, death, or until 12 months
Measure: Mean (95% Confidence Interval); unit: percentage of event free participants
Groups:
- Group 1: In Group 1, PCI-32765 420 mg PO daily was administered daily for 1 cycle (28 days) before the start of ofatumumab IV dosing
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 27 | 20 | 24
percentage of event free participants | 88.7 [69.0 to 96.2] | 85.0 [60.4 to 94.9] | 75.0 [52.6 to 87.9]

4. Primary Outcome: Safety During Dose-Limiting Toxicity (DLT) Observation Period
Description: Number of dose-limiting toxicities observed in the first 6 participants enrolled in treatment Groups 1 and 2
Time Frame: 56 days for Group 1 and 28 days for Group 2
Measure: Number; unit: participants who experienced DLT
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 6 | 6
participants who experienced DLT | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study treatment to within 30 days of last dose or until study closure
Arm/Group | Group 1 | Group 2 | Group 3
Serious Adverse Events (participants affected / at risk) | 12/27 | 9/20 | 10/24
Other Adverse Events (participants affected / at risk) | 27/27 | 20/20 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=27) | Group 2 (N=20) | Group 3 (N=24)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 4 | 3 | 4
Cellulitis (Infections and infestations) | 1 | 0 | 2
Pneumonia fungal (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Pneumonia pseudomonas aeruginosa (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Richter's syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=27) | Group 2 (N=20) | Group 3 (N=24)
Neutropenia (Blood and lymphatic system disorders) | 4 | 5 | 3
Anaemia (Blood and lymphatic system disorders) | 7 | 2 | 2
Increased tendency to bruise (Blood and lymphatic system disorders) | 10 | 5 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 2
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 3 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0 | 2
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1
Haematotympanum (Ear and labyrinth disorders) | 0 | 1 | 0
Motion sickness (Ear and labyrinth disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 3
Eye haemorrhage (Eye disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 1 | 1 | 1
Vision blurred (Eye disorders) | 0 | 3 | 1
Cataract (Eye disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 4 | 0 | 0
Intraocular haematoma (Eye disorders) | 0 | 1 | 0
Iridocyclitis (Eye disorders) | 1 | 0 | 0
Iris adhesions (Eye disorders) | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 1 | 0
Photophobia (Eye disorders) | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 18 | 16 | 16
Stomatitis (Gastrointestinal disorders) | 11 | 9 | 7
Nausea (Gastrointestinal disorders) | 5 | 6 | 6
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 2
Dry mouth (Gastrointestinal disorders) | 3 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 4 | 2
Oral pain (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 2 | 0 | 1
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 3 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 1 | 0
Tongue blistering (Gastrointestinal disorders) | 1 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 1 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3 | 0
Oedema peripheral (General disorders) | 7 | 2 | 4
Chills (General disorders) | 2 | 0 | 3
Pain (General disorders) | 1 | 0 | 2
Chest discomfort (General disorders) | 1 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 13 | 1 | 1
Localised oedema (General disorders) | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0
Axillary pain (General disorders) | 1 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 0
Catheter site rash (General disorders) | 1 | 0 | 0
Injection site bruising (General disorders) | 1 | 0 | 0
Irritability (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0
Temperature intolerance (General disorders) | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0
Portal hypertension (Hepatobiliary disorders) | 1 | 0 | 0
Sarcoidosis (Immune system disorders) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 7 | 8 | 5
Sinusitis (Infections and infestations) | 6 | 2 | 3
Urinary tract infection (Infections and infestations) | 5 | 2 | 3
Bronchitis (Infections and infestations) | 2 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1
Ear infection (Infections and infestations) | 1 | 1 | 1
Infection (Infections and infestations) | 0 | 0 | 1
Nasal abscess (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 2 | 1
Pneumonia fungal (Infections and infestations) | 0 | 0 | 1
Eye infection (Infections and infestations) | 1 | 2 | 0
Eye infection toxoplasmal (Infections and infestations) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 2 | 1 | 0
Furuncle (Infections and infestations) | 1 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 4 | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Infected bites (Infections and infestations) | 1 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 6 | 3 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 2 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Tinea infection (Infections and infestations) | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 9 | 14 | 9
Contusion (Injury, poisoning and procedural complications) | 9 | 8 | 3
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 5 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 3 | 0 | 0
Periorbital contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 | 0 | 0
Skin wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 2 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0
Grip strength decreased (Investigations) | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Weight increased (Investigations) | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 2 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 2 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 3 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 4 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 11 | 8 | 12
Headache (Nervous system disorders) | 2 | 1 | 3
Dizziness (Nervous system disorders) | 4 | 4 | 1
Dizziness postural (Nervous system disorders) | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 4 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 1
Confusional state (Psychiatric disorders) | 4 | 0 | 0
Insomnia (Psychiatric disorders) | 5 | 6 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Renal mass (Renal and urinary disorders) | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Vocal cord cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 6 | 5 | 6
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Blood blister (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 3 | 2 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 5 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Flushing (Vascular disorders) | 4 | 2 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 2 | 3 | 0
Peripheral artery aneurysm (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No